CLINICAL TRIAL: NCT01267578
Title: Phase II Multicenter Trial of Peptide Vaccination Therapy Using Novel Cancer Testis Antigens (STF-II) for Locally Advanced, Recurrent, or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: Peptide Vaccination in Treating Patients With Esophageal Cancer (STF-II)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Yamanashi (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: First Department of Surgery, University of Yamanashi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMU-03
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Esophageal Cancer
Keywords: Epitope peptide, CTL, Esophageal cancer, Vaccination
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peptide vaccination (Experimental)
  Interventions: Biological: vaccination

INTERVENTIONS:
Biological: vaccination — Biological/Vaccine: URLC10, CDCA1, and KOC1 peptides

SUMMARY:
The purpose of this study is to evaluate overall survival and immunological monitoring for peptide vaccination therapy using novel cancer testis antigens (STF-II) for locally advanced, recurrent, or metastatic esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
The phase II multicenter trial of vaccination study using peptides derived from URLC10, CDCA1, and KOC1 for locally advanced, recurrent or metastatic esophageal squamous cell carcinoma (ESCC) who had failed for the standard therapy are performed to evaluate the survival benefit of the cancer vaccination.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

1. Locally advanced, recurrent or metastatic esophageal squamous cell carcinoma who had failed for the standard therapy

PATIENTS CHARACTERISTICS

1. ECOG performance status 0-2
2. Age≧20 years, 80≦years
3. WBC≥ 2,000/mm³ Platelet count ≥ 75,000/mm³ Total bilirubin ≤ 2.0 x the institutional normal upper limits AST, ALT, ALP ≤ 2.5 x the institutional normal upper limits Creatinine ≤ 1.5 x the institutional normal upper limits
4. No therapy 4 weeks prior to the initiation of the trial
5. Able and willing to give valid written informed consent -

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Serious bleeding disorder
4. Serious infections requiring antibiotics
5. Concomitant treatment with steroids or immunosuppressing agent
6. Decision of unsuitableness by principal investigator or physician-in-charge -

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | death from start of treatment

SECONDARY OUTCOMES:
CTL response | CTL response after 5 round vaccination
DTH response | Skin reaction after 5 round vaccination
Progression free survival | time from start of vaccination until disease progreesion

CONTACTS AND LOCATIONS:
Overall Officials: Koji Kono, PhD, MD, Principal Investigator — University of Yamanashi, First Department of Surgery
Locations (1):
- University of Yamanashi, First Department of Surgery, Chūō, Yamanashi, Japan

REFERENCES:
- [Background] 1. Okabe H, Satoh S, Kato T, et al. Genome-wide analysis of gene expression in human hepatocellular carcinomas using cDNA microarray: identification of genes involved in viral carcinogenesis and tumor progression. Cancer Res 2001; 61: 2129-37. 2 Lin YM, Furukawa Y, Tsunoda T, Yue CT, Yang KC, Nakamura Y. Molecular diagnosis of colorectal tumors by expression profiles of 50 genes expressed differentially in adenomas and carcinomas. Oncogene 2002; 21: 4120-28. 3. Hasegawa S, Furukawa Y, Li M, et al. Genome-wide analysis of gene expression in intestinal-type gastric cancers using a complementary DNA microarray representing 23,040 genes. Cancer Res 2002; 62: 7012-17. 4. Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci 2007; 98: 1803-8. 5. Ishikawa N, Takano A, Yasui W, et al. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res 2007; 67: 11601-11. 6. Yoshiki Mizukami, Koji Kono, Yataro Daigo, et al. Detection of novel Cancer-Testis antigen-specific T-cell responses in TIL, regional lymph nodes and PBL in patients with esophageal squamous cell carcinoma. Cancer Science 2008 ;99:1448-54 6. Koji Kono, Yoshiki Mizukami, Yataro Daigo, Atsushi Takano, Ken Masuda, Koji Yoshida, Takuya Tsunoda, Yoshihiko Kawaguchi, Yusuke Nakamura, and Hideki Fujii. Vaccination with Multiple Peptides derived from Novel Cancer-Testis Antigens Can Induce Specific T-Cell Responses and Clinical Responses in Advanced Esophageal cancer. Cancer Sci. 2009;100:1502-9.